CLINICAL TRIAL: NCT06964126
Title: "Psycho-Social Effects of Gardening Activities in the Elderly: An Investigation on Self-Esteem and Life Satisfaction
Brief Title: Psycho-Social Effects of Gardening Activities in the Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: Gardening activities
Record Dates: First submitted 2025-04-24; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Life Satisfaction; Self Esteem
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gardening Activities Group (Experimental): Gardening activities will be applied to this group.In the study, the elderly individuals in the experimental group will have a total of 8 sessions of gardening activities once a week (on Thursday) for 2 months. Before the gardening activities, the garden and environment will be prepared by the researcher, the elderly individuals will be informed about the day's activities and, if necessary, videos about the activities will be watched and photographs related to the sessions will be shown.
  Interventions: Other: Horticulture activities
- Control Group (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Other: Horticulture activities — In the study, the elderly individuals in the experimental group will have a total of 8 sessions of gardening activities once a week (on Thursday) for 2 months. Before the gardening activities, the garden and environment will be prepared by the researcher, the elderly individuals will be informed about the day's activities and, if necessary, videos about the activities will be watched and photographs related to the sessions will be shown.
  Arms: Gardening Activities Group

SUMMARY:
In this study titled "Psycho-Social Effects of Gardening Activities in the Elderly: A Study on Self-Esteem and Life Satisfaction", the elderly will be divided into two groups as experimental and control groups. Participants will be randomly assigned to the groups. No intervention will be made to the patients in the control group. Gardening activities will be performed on the patients in the experimental group as of April. The following questions will be answered in this study;

Do gardening activities affect the self-esteem level of the elderly? Do gardening activities affect the life satisfaction level of the elderly?

DETAILED DESCRIPTION:
In this study titled "Psycho-Social Effects of Gardening Activities in the Elderly: A Study on Self-Esteem and Life Satisfaction", the elderly will be divided into two groups as experimental and control groups. Participants will be randomly assigned to the groups. No intervention will be made to the patients in the control group. Gardening activities will be performed on the patients in the experimental group as of April. The study is very important as it is the first of its kind in the literature. In addition, it is thought that the results of this study will contribute scientifically to psychiatric nurses who care for elderly individuals and to the literature in the field of nursing. Data will be collected using the "Life Satisfaction Scale" and the "Rosenberg Self-Esteem Scale Short Form Scale".

The following questions will be answered in this study; Do gardening activities affect the self-esteem level of the elderly? Do gardening activities affect the life satisfaction level of the elderly?

ELIGIBILITY:
Inclusion Criteria:

* The elderly who have a Standardized Mini Mental Test score of 24 and above,
* Do not have vision or hearing loss that may prevent gardening activities,
* Are open to communication and cooperation,
* Volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Having a communication problem
* Having attended a gardening training in the last 6 months
* Having a physical illness that would prevent gardening activities
* Having a psychiatric illness that would prevent gardening activities will be excluded from the study.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Life Satisfaction | 2 months
  Scale score average; This scale, consisting of 5 items, has a 7-point Likert-type rating ("1" Strongly disagree - "7" Strongly agree). High scores indicate high levels of life satisfaction. The highest score that can be obtained from the scale is 35; the lowest score is 5.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Çapar, Speciaalist, Study Director — http://www.agin.gov.tr/ilce-toplum-sagligi-merkezi
Locations (1):
- Ağın Community Health Center, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No